CLINICAL TRIAL: NCT03789825
Title: Screening for Liver Fibrosis. A Population-based Study in European Countries. The ''LiverScreen'' Project.
Brief Title: Population-based Study in Screening for Liver Fibrosis
Acronym: LiverScreen
Status: Completed | Type: Observational
Sponsor: Judit Pich Martínez (Other)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Other Study IDs: LiverScreen
Record Dates: First submitted 2018-11-14; First posted 2018-12-31 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum specimens will be retained in a repository
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study to assess the prevalence of significant liver fibrosis in general population using Transient Elastography

DETAILED DESCRIPTION:
This is a population-based study. Subjects will attend a primary care center where a physical examination, general blood test and transient elastography will be carried out. Only the group of patients with high-risk for liver fibrosis will be evaluated in a second visit at the University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Able to give informed consent

Exclusion Criteria:

* Previously known chronic liver disease (including cholestasis). Patients with already known liver steatosis but no diagnosis of liver fibrosis or cirrhosis can be included
* Subjects with mental incapacity, language barrier, insufficient social support or any other reason considered by the investigator precluding adequate understanding or cooperation in the study
* Subjects with a history of current malignancy including solid tumors and hematologic disorders
* Subjects with significant extrahepatic disease that may impair short-term prognosis (including congestive heart failure New York Heart Association Grade IV, COPD GOLD >3)
* Subjects with kidney disease (serum creatinine >3mg/dL or under renal replacement therapy)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population above 40 years
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
% of subjects with Liver stiffness measurement by Transient Elastography >=8 kPa at any visit | Through study completion, an average of 24 months
  Percentage of subjects with Liver stiffness measurement by Transient Elastography ≥ 8 kPa at any visit, either with M or XL probe, in general population.

SECONDARY OUTCOMES:
% of subjects with Liver stiffness measurement by Transient Elastography >=8 kPa in the subgroup of patients with risk factors for chronic liver disease at visit 1 or 2 | Through study completion, an average of 24 months
  Percentage of subjects with Liver stiffness measurement by Transient Elastography ≥ 8 kPa, either with M or XL probe, in the subgroup of patients with risk factors for chronic liver disease at visit 1 and/or 2.
Comparison of liver fibrosis diagnosis accuracy between Transient Elastography and fibrosis scores | Through study completion, an average of 24 months
  Comparison of liver fibrosis diagnosis accuracy between Transient Elastography and fibrosis scores (including NAFLD fibrosis score, FIB-4, Forms index and APRI score) for the diagnosis of liver fibrosis in general population and in the subgroup of patients with risk factors for chronic liver disease at visit 1 and 2.
Comparison of liver fibrosis diagnosis accuracy between Transient Elastography, fibrosis scores and liver biopsy | Through study completion, an average of 24 months
  Comparison of liver fibrosis diagnosis accuracy between Transient Elastography, fibrosis scores and liver biopsy for the diagnosis of liver fibrosis in general population and in the subgroup of patients with risk factors for chronic liver disease, in patients with liver biopsy available at visit 2.
% of subjects with CAP ≥250 dB/m | Through study completion, an average of 24 months
  Percentage of subjects with CAP ≥250 dB/m, either with M or XL probe, in general population and in the subgroup of patients with risk factors for chronic liver disease at visit 1 and/or 2
Comparison of liver steatosis diagnosis accuracy between CAP and steatosis scores | Through study completion, an average of 24 months
  Comparison of liver steatosis diagnosis accuracy between CAP and steatosis scores (including FLI, HIS, LAP, ION and NAFLD-LFS) for the diagnosis of liver steatosis in general population and in the subgroup of patients with risk factors for chronic liver disease at visit 1 and 2.
Comparison of liver steatosis diagnosis accuracy between CAP, steatosis scores and liver biopsy | Through study completion, an average of 24 months
  Comparison of liver steatosis diagnosis accuracy between CAP, steatosis scores (including FLI, HIS, LAP, ION and NAFLD-LFS) and liver biopsy for the diagnosis of liver steatosis in general population and in the subgroup of patients with risk factors for chronic liver disease, in patients with liver biopsy available (at visit 2).
Comparison of liver steatosis diagnosis accuracy between CAP and abdominal ultrasound | Through study completion, an average of 24 months
  Comparison of liver steatosis diagnosis accuracy between CAP and abdominal ultrasound for the diagnosis of liver steatosis in general population and in the subgroup of patients with risk factors for chronic liver disease, in patients with abdominal ultrasound available at visit 2.
Comparison of values obtained with M and XL probes in the assessment of LSM and CAP via TE | Through study completion, an average of 24 months
  Comparison of values obtained with M and XL probes in the assessment of LSM and CAP via TE at visit 2.
Cost-effectiveness of a liver fibrosis screening program for liver fibrosis detection in general population | Through study completion, an average of 24 months
  Cost-effectiveness of a liver fibrosis screening program for liver fibrosis detection in general population and in the subgroup of patients with risk factors for chronic liver disease. Direct and indirect cost savings of early detection of liver fibrosis in subjects with risk factors for chronic liver diseases.
Percentage of failure rate for stiffness and steatosis measurements within TE examination | Through study completion, an average of 24 months
  Percentage of failure rate for stiffness and steatosis measurements within TE examination at visit 1 and 2.
Percentage of patients with procedure related adverse events and serious adverse events | Through study completion, an average of 24 months
  Percentage of patients with procedure related adverse events (adverse events related to TE and liver biopsy) and serious adverse events during all the duration of the study.
Percentage of patients with changes in lifestyle habits | Through study completion, an average of 24 months
  Percentage of patients with changes in lifestyle habits

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, MD, Study Chair — Fundacion Clinic per a la Recerca Biomédica
Locations (45):
- Croatia (2):
  - Dubrava Hospital, Zagreb
  - Poliklinika Croatia, Zagreb
- Odense University Hospital, Odense, Denmark
- France (4):
  - Centre de santé Municipal Etienne Gatineau-Sailliant de Genevilliers, Gennevilliers
  - Centre de Recherche Clinique - CRC, Paris
  - Hospital Avicenne, Paris
  - Hospital Beaujon, Paris
- Germany (5):
  - Homburg Hospital, Homburg
  - Altstadtpraxis, Mainz
  - Mainz Hospital, Mainz
  - Praxis Mombach, Mainz
  - MVZ Dres.Schneider Kaiserslautern, Rodenbach
- Italy (2):
  - Medicina Di gruppo di montagnana, Padua
  - Vigonza Medica, Padua
- Medical Center Rotterdam, Rotterdam, Netherlands
- F. D. Roosevelt Univ. Hospital, Banská Bystrica, Slovakia
- Spain (21):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - SEAT, Martorell, Barcelona
  - CAP II El Maresme, Mataró, Barcelona
  - CAP II Santa Coloma de Gramanet, Santa Coloma de Gramenet, Barcelona
  - CAP La Florida, Santa Perpètua de Mogoda, Barcelona
  - CAP Barceloneta, Barcelona
  - Hospital del Mar, Barcelona
  - CAP Bordeta-Magòria, Barcelona
  - CAP Río de Janeiro, Barcelona
  - CAP Ciutat Meridiana, Barcelona
  - CAP Sant Rafael, Barcelona
  - Hospital Universirati Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - CAP Adrià, Barcelona
  - CAP Besos, Barcelona
  - CAP La Marina, Barcelona
  - CAP Numància, Barcelona
  - CAP Vila de Gracia, Barcelona
  - CAP Vila Olimpica, Barcelona
  - Hospital Gregorio Marañon, Madrid
  - CAP La Llantia, Mataró
- United Kingdom (8):
  - Oak Lodge Medical Centre, Edgware
  - Royal Free Hospital, London
  - James Wigg, London
  - Mild May, London
  - Oakleigh park, London
  - St Andrews Medical Practice, London
  - Nottingham University Hospital, Nottingham
  - King's Mill Hospital, Sutton in Ashfield

REFERENCES:
- [Derived] Graupera I, Thiele M, Ma AT, Serra-Burriel M, Pich J, Fabrellas N, Caballeria L, de Knegt RJ, Grgurevic I, Reichert M, Roulot D, Schattenberg JM, Pericas JM, Angeli P, Tsochatzis EA, Guha IN, Garcia-Retortillo M, Morillas RM, Hernandez R, Hoyo J, Fuentes M, Madir A, Juanola A, Soria A, Juan M, Carol M, Diaz A, Detlefsen S, Toran P, Pera G, Fournier C, Llorca A, Newsome PN, Manns M, de Koning HJ, Serra-Burriel F, Cucchietti F, Arslanow A, Korenjak M, van Kleef L, Falco JL, Kamath PS, Karlsen TH, Castera L, Lammert F, Krag A, Gines P; LiverScreen Consortium investigators. LiverScreen project: study protocol for screening for liver fibrosis in the general population in European countries. BMC Public Health. 2022 Jul 19;22(1):1385. doi: 10.1186/s12889-022-13724-6. PMID 35854275